CLINICAL TRIAL: NCT06348888
Title: A Phase 1 Open Label, Two-arm, Fixed Sequence, Crossover Study to Investigate the Effects of Itraconazole and Carbamazepine on the Pharmacokinetics of BAY 2927088 in Healthy Participants
Brief Title: A Study to Learn About How Itraconazole and Carbamazepine Affect the Level of BAY2927088 in the Blood When These Drugs Are Taken Together by Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22250
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Advanced Non-small Cell Lung Cancer; EGFR Mutation; HER2 Mutation; Healthy Volunteers
Keywords: HER2 (Human epidermal growth factor receptor 2); EGFR (Epidermal growth factor receptor); NSCLC (Non-small cell lung cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Itraconazole; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAY2927088 + Itraconazole (ITZ) (Experimental): Participant will receive single dose BAY2927088 on Days 1 and 8, will receive itraconazole daily from Day 5 to Day 11.
  Interventions: Drug: BAY2927088; Drug: Itraconazole
- BAY2927088 + Carbamazepine (CBZ) (Experimental): Participant will receive BAY2927088 single dose on Days 1 and 14, will receive carbamazepine daily from Day 3 to Day 15.
  Interventions: Drug: BAY2927088; Drug: Carbamazepine

INTERVENTIONS:
Drug: BAY2927088 — Oral
Drug: Itraconazole — Capsule, 100 mg, oral.
  Arms: BAY2927088 + Itraconazole (ITZ)
Drug: Carbamazepine — Tablet, 100 mg, 200mg and 300mg, oral.
  Arms: BAY2927088 + Carbamazepine (CBZ)

SUMMARY:
Researchers are looking for a better way to treat people who have advanced non-small cell lung cancer (NSCLC) with specific genetic changes called EGFR and HER2 mutations.

Advanced NSCLC refers to a type of lung cancer that has spread from the lungs to nearby tissues or other body parts. People with advanced NSCLC may have changes in certain proteins like EGFR and HER2, that cause uncontrolled cell growth and increased spread of cancer.

In this study, participants will be healthy and will not benefit from taking the study treatment, BAY2927088. However, the study will provide information about how to test BAY2927088 in future studies with people who have advanced NSCLC with EGFR or HER2 mutations.

BAY2927088 is under development for the treatment of advanced NSCLC with EGFR or HER2 mutations. It is expected to work against these changed proteins, which might slow down the spread of cancer.

BAY2927088 is broken down by an enzyme called CYP3A4 inside the body. Itraconazole is a drug that inhibits the activity of CYP3A4 while carbamazepine is a drug that enhances the activity of CYP3A4. Giving these drugs together will allow researchers to learn how the blood levels of BAY2927088 change when the CYP3A4 activity is inhibited or enhanced.

The main purpose of this study is to find out how itraconazole and carbamazepine may affect the blood levels of BAY2927088. For this, researchers will measure the following for BAY2927088 when it is given with and without itraconazole and carbamazepine

* Area under the curve (AUC): a measure of the total amount of BAY2927088 in participants' blood over time
* Maximum observed concentration (Cmax): the highest amount of BAY2927088 in participants' blood

The study will have 2 treatment groups.

In Group 1, participants will take:

* BAY2927088 as a single dose on Days 1 and 8.
* Itraconazole once daily on Days 5 to 11.

In Group 2, participants will take:

* BAY2927088 as a single dose on Days 1 and 14.
* Different doses of carbamazepine two times a day on Days 3 to 15. Participants will be in this study for about 7 weeks in Group 1 and 8 weeks in Group 2.

Participants will visit the study clinic:

* at least once, 2 to 28 days before the treatment starts in both groups, to confirm they can take part in this study
* on Day 1, and will stay at the clinic until Day 12 in Group 1 and Day 16 in Group 2
* once, 7 to 10 days later from last dose of BAY2927088 in both groups, for a health check up

During the study, the doctors and their study team will:

* perform physical examinations
* collect blood samples from the participants to measure the levels of BAY2927088
* check participants' health by performing tests such as blood and urine tests, and checking heart health using an electrocardiogram (ECG)
* ask the participants questions about how they are feeling and what adverse events they are having An adverse event is any medical problem that a participant has during a study. The study doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent as described in protocol, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF), and in this protocol.
* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, laboratory tests, physical, and cardiac examination.
* Participant is a nonsmoker who has not used tobacco- or nicotine- containing products (eg., nicotine patch) for at least 6 months before administration of the first study intervention.
* Body mass index (BMI) within the range 18.0 to 30 kg/m2 (inclusive) at screening, with bodyweight above/equal to 50 kg.
* Female, of non childbearing potential only. Females must not be pregnant or breastfeeding, and must be documented as a woman of nonchildbearing potential. A negative pregnancy test is required.
* Male study participants of reproductive potential must agree to use adequate contraception when sexually active. From signing of the ICF until at least 3 months after the last dose of study intervention, and refrain from sperm donation during study intervention and for 6 months after the last dose of study intervention.
* Participant must be willing to comply with dietary and fluid requirements during the study period (including abstaining from alcohol use).

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g., liver diseases, heart diseases, gastrointestinal diseases, interstitial lung disease, renal diseases), central nervous system (for example seizures) or other organs (e.g., diabetes mellitus).
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study intervention will not be normal.
* Febrile illness within 4 weeks prior to admission to the clinic.
* Any relevant diseases within 4 weeks prior to the first study intervention administration as judged by the investigator.
* A medical history of risk factors for Torsades de pointes (e.g., family history of long QT syndrome) or other clinically significant arrhythmias as judged by the investigator.
* Known severe allergies, allergies requiring therapy with corticosteroids, significant non-allergic drug reactions, or (multiple) drug allergies (excluding seasonal allergies such as non-severe hay fever that are asymptomatic and untreated during the time of study conduct).
* Known history of hypersensitivity (or known allergic reaction) to BAY2927088 related compounds, or any components of the formulation, itraconazole or carbamazepine (HLA-A 31:01 or HLA-B 15:02 allele for Arm 2 only)
* History of known or suspected malignant tumors.
* Participants with any type of ongoing psychiatric disorder, especially any mood disorders including medical history with suicidal ideation and/or suicide attempts, which may disable the participant to consent.
* History of clinically relevant depression, or suicidal ideation or behavior.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
AUC of BAY2927088 with and without itraconazole | Pre-dose of Day 1, multiple post-dose time points of Days 1-5, pre-dose of Day 8, multiple post-dose time points of Days 8-12
Cmax of BAY2927088 with and without itraconazole | Pre-dose of Day 1, multiple post-dose time points of Days 1-5, pre-dose of Day 8, multiple post-dose time points of Days 8-12
AUC of BAY2927088 with and without carbamazepine | Pre-dose of Day 1, multiple post-dose time points of Days 1-3; pre-dose of Day 14, multiple post-dose time points of Days 14-16
Cmax of BAY2927088 with and without carbamazepine | Pre-dose of Day 1, multiple post-dose time points of Days 1-3; pre-dose of Day 14, multiple post-dose time points of Days 14-16

SECONDARY OUTCOMES:
Number of participants with TEAEs | After the first administration of study intervention up to 7 days after the last administration of study intervention.
Severity of TEAEs | After the first administration of study intervention up to 7 days after the last administration of study intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Baltimore - Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — http://clinicaltrials.bayer.com/study/22250